CLINICAL TRIAL: NCT05671757
Title: Targeting CD38 With Daratumumab in Primary Antiphospholipid Syndrome: A Phase 1b Dose Escalation Safety Trial (ITN093AI)
Brief Title: Daratumumab in Primary Antiphospholipid Syndrome
Acronym: DARE-APS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN093AI
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Autoimmune Disorders
Keywords: Daratumumab; Anti-Phospholipid Syndrome
MeSH Terms: conditions — Autoimmune Diseases; Antiphospholipid Syndrome | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 4 mg/kg Cohort (Experimental): This cohort will receive intravenous (IV) administration of 4 mg/kg daratumumab administered weekly for 8 doses (weeks 0 through 7). Post-treatment follow-up visits will occur at weeks 9, 12, 18, 24, 36, and 48
  Interventions: Biological: Daratumumab
- 8 mg/kg Cohort (Experimental): This cohort will receive intravenous (IV) administration of 8 mg/kg daratumumab administered weekly for 8 doses (weeks 0 through 7). Post-treatment follow-up visits will occur at weeks 9, 12, 18, 24, 36, and 48
  Interventions: Biological: Daratumumab
- 16 mg/kg Cohort (Experimental): This cohort will receive intravenous (IV) administration of 16 mg/kg daratumumab administered weekly for 8 doses (weeks 0 through 7). Post-treatment follow-up visits will occur at weeks 9, 12, 18, 24, 36, and 48
  Interventions: Biological: Daratumumab

INTERVENTIONS:
Biological: Daratumumab — Participants will receive 4 mg/kg of intravenous (IV) daratumumab administered weekly for 8 doses (weeks 0 through 7). Post-treatment follow-up visits will occur at weeks 9, 12, 18, 24, 36, and 48
  Other Names: DARZALEX; DARZALEX®
  Arms: 4 mg/kg Cohort
Biological: Daratumumab — Participants will receive 4-8 mg/kg of intravenous (IV) daratumumab administered weekly for 8 doses (weeks 0 through 7). Post-treatment follow-up visits will occur at weeks 9, 12, 18, 24, 36, and 48
  Other Names: DARZALEX; DARZALEX®
  Arms: 8 mg/kg Cohort
Biological: Daratumumab — Participants will receive 4-16 mg/kg of intravenous (IV) daratumumab administered weekly for 8 doses (weeks 0 through 7). Post-treatment follow-up visits will occur at weeks 9, 12, 18, 24, 36, and 48
  Other Names: DARZALEX; DARZALEX®
  Arms: 16 mg/kg Cohort

SUMMARY:
The purpose of this study is to see if the study medication, daratumumab, is safe to treat individuals with Anti-Phospholipid Syndrome (APS).

Three daratumumab dosing cohorts are planned with up to six participants in each dosing cohort with the potential to enroll an additional 4 subjects in the highest safe dose (HSD) cohort, for a total of up to 22 participants. The dosing cohorts are: 4 mg/kg, 8 mg/kg, and 16 mg/kg. Each cohort will receive intravenous (IV) administration of daratumumab according to the following schedule, for a total of 8 doses.

The primary objective is to determine the safety of daratumumab in APS defined as Dose Limiting Toxicities (DLTs) occurring during the dose escalation phase.

DETAILED DESCRIPTION:
The trial is a phase 1b open-label study of daratumumab in participants with APS.

The study design is a modification of the 3 + 3 dose escalation scheme. Three daratumumab dose cohorts are planned: 4 mg/kg, 8 mg/kg, and 16 mg/kg of intravenous (IV) daratumumab administered weekly for 8 doses (weeks 0 through 7). Post-treatment follow-up visits will occur at weeks 9, 12, 18, 24, 36, and 48.

Dose Escalation Phase Dose escalation will proceed according to safety criteria (Dose Limiting Toxicity, DLT) and efficacy criteria (antiphospholipid antibody negativity). An independent safety committee will review the data and approve escalation to the next dose.

The Highest Safe Dose (HSD) is the highest administered dose at which ≤ 1/6 participants experiences a DLT at or prior to week 9.

Expansion Phase Four additional participants will be enrolled and treated at the HSD weekly for 8 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 70 years of age, inclusive.
2. The completion of the following vaccinations at least 14 days prior to Visit 0:

   1. At least one dose of the most recently updated COVID-19 vaccine, and
   2. At least one dose of the herpes zoster vaccination series, and
   3. Current seasonal influenza vaccine, if available.
3. History of APS according to the updated 2006 Sapporo classification criteria, including at least one of the following:

   a. Arterial thrombosis, except transient ischemic attack, confirmed by objective validated criteria such as imaging, or b. Venous thrombosis, except superficial thrombophlebitis, confirmed by objective validated criteria such as imaging, or c. Pregnancy morbidity, based on the updated 2006 Sapporo APS classification criteria, or d. Microvascular APS, with at least one of the following: i. Renal biopsy documentation of aPL-associated nephropathy, or ii. Lung biopsy or bronchoalveolar lavage documentation of diffuse alveolar hemorrhage (DAH), or iii. Skin biopsy documentation of livedoid vasculopathy.
4. History of triple positive aPL within the prior 5 years and at least 12 weeks prior to enrollment, including all of the following:

   1. aCL IgG level > Upper Limit of Normal (ULN), and
   2. aβ2GPI IgG level > ULN, and
   3. Positive LA test.
5. Confirmation of triple positive aPL at screening, including all of the following:

   1. aCL IgG level ≥ 40 GPL, and
   2. aβ2GPI IgG level ≥ 40 SGU, and
   3. Positive LA test.
6. Undergoing anticoagulation with warfarin or low molecular weight heparin (LMWH), if there is a history of arterial or venous thrombosis.

Exclusion Criteria:

1. Inability or unwillingness to give written informed consent.
2. Inability or unwillingness to comply with study protocol.
3. Systemic autoimmune diseases other than APS, including but not limited to:

   1. Systemic lupus erythematosus (SLE) meeting the EULAR/ACR classification criteria.
   2. Rheumatoid arthritis meeting the ACR/EULAR classification criteria.
   3. Small, medium, and large vessel vasculitis meeting ACR classification criteria.
4. Catastrophic APS classification within the prior 90 days.
5. Acute arterial or venous thrombosis within the prior 30 days.
6. Use of the following medications:

   1. Any prior treatment with CD38 targeting monoclonal antibodies, including daratumumab or isatuximab-irfc.
   2. The following within the prior 30 days:

   i. Corticosteroids > 10 mg/day prednisone or equivalent. ii. Direct oral anticoagulants (DOACs). iii. Live attenuated vaccines. iv. IVIG or other supplemental immunoglobulin. c. Azathioprine, methotrexate, mycophenolate mofetil, mycophenolate sodium, lefluonomide, or calcineurin inhibitors within the prior 90 days.

   d. Cyclophosphamide within the prior 90 days. e. Immunomodulatory or immunosuppressive biologic agents, including belimumab, within the prior 90 days or 5 half-lives, whichever is greater.

   f. Investigational agents within the prior 90 days or 5 half-lives, whichever is greater, except for COVID-19 vaccines and medications for prevention or treatment of COVID-19 per FDA Emergency Use Authorization (EUA).

   g. Biologic B cell depleting agents including rituximab with any of the following: i. Treatment within the prior 180 days, or ii. CD19+ absolute count < 40/ μl, or iii. Serum IgG <500 mg/dL.
7. Plasma exchange within the prior 90 days.
8. Hemodialysis within the prior 90 days.
9. Major surgical procedure within the prior 60 days.
10. Known allergy, hypersensitivity, or intolerance to boron, malitol, sorbitol, corticosteroids, monoclonal antibodies including daratumumab, human proteins, or their excipients.
11. Allergy, intolerance, or contraindication to acyclovir, valacyclovir, and famciclovir.
12. Active or chronic infection, including the following:

    1. Active bacterial, viral, fungal, or opportunistic infection.
    2. Chronic infection requiring suppressive antibiotic treatment.
    3. Intravenous antibiotics or hospitalization for infection within the prior 30 days.
    4. Evidence of current or prior Mycobacterium tuberculosis infection.
    5. Human immunodeficiency virus (HIV).
    6. Current or prior infection with hepatitis B virus (HBV).
    7. Current or prior infection with hepatitis C virus (HCV), except adequately treated HCV with sustained virologic response ≥ 12 weeks.
    8. History of recurrent herpes zoster, or history of herpes zoster ophthalmicus, disseminated herpes zoster, or disseminated herpes simplex.
13. The following laboratory abnormalities:

    ITN093AI: DARE-APS Version 3.0 September 12, 2023 Daratumumab in Primary Antiphospholipid Syndrome
    1. Absolute neutrophil count < 1500/mm3.
    2. Platelets < 100,000/mm3.
    3. Hemoglobin (Hgb) < 10 g/dL.
    4. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase > 2x the Upper Limit of Normal (ULN).
    5. Total bilirubin > 2x ULN, except in the case of congenital bilirubinemia then direct bilirubin > 2x ULN.
    6. eGFR < 45 ml/min/1.73 m2.
14. History of primary immunodeficiency.
15. History of solid organ or hematopoietic stem cell transplantation.
16. Comorbidities requiring systemic corticosteroid therapy, including those which have required three or more courses of systemic corticosteroids within the 12 months prior to Visit 0.
17. Any of the following conditions with FEV1 < 70% predicted within the prior 90 days:

    1. Asthma.
    2. Chronic obstructive pulmonary disease (COPD).
    3. DAH.
18. Pulmonary hypertension.
19. Adrenal insufficiency.
20. Poorly controlled diabetes mellitus defined as hemoglobin A1c (HbA1c) ≥ 8.0%.
21. Concomitant malignancy or history of malignancy, except adequately treated or excised nonmetastatic squamous cell carcinoma, basal cell skin carcinoma, or cervical carcinoma in situ.
22. Clinically significant cardiac disease, including but not limited to:

    1. Myocardial infarction within the prior 6 months, or
    2. Unstable or uncontrolled disease or condition related to or affecting cardiac function, including but not limited to:

    i. Unstable angina, or ii. Congestive heart failure, New York Heart Association Class II-IV, or iii. Uncontrolled cardiac arrhythmia.
23. Current diagnosed mental illness or current diagnosed or self-reported drug or alcohol abuse which, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
24. Severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, or neurological disease.
25. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or may impact the quality or interpretation of the data obtained from the study.
26. Lack of peripheral venous access.
27. Pregnancy, or planning a pregnancy during the 48 week study duration.
28. Breast-feeding.
29. Unwillingness to use medically acceptable non-prothrombotic contraception if of reproductive potential and engaging in sexual activity that could lead to pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants in the dose escalation phase with at least one Dose Limiting Toxicity (DLT) | At or before week 9
  Proportions will be estimated by dose cohort with 95% confidence intervals derived using the Clopper-Pearson exact method

SECONDARY OUTCOMES:
The proportion of Grade 2 or higher adverse event (AEs) and serious adverse events (SAEs) related to daratumumab | At or before weeks 9, 24, and 48
  The proportion of participants who experience at least one event will be estimated by dosing level with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with the following Grade 3 or higher adverse events (AEs) related to daratumumab | At or before weeks 9, 24, and 48.
  Adverse events including:
  1. Infusion reaction
  2. Neutropenia
  3. Thrombocytopenia
  4. Infection
The proportion of participants with negative Lupus Anticoagulant (LA) test | At week 9
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with at least 50% reduction in Anticardiolipin antibodies Immunoglobulin G (aCL IgG) | At week 9 compared to week 0
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with at least 50% reduction in Anti-beta2-glycoprotein test Immunoglobulin G (abeta2GPI IgG) levels | At week 9 compared to week 0
The proportion of participants with at least 50% reduction in Anticardiolipin antibodies Immunoglobulin G (aCL IgG) levels | At week 24 compared to week 0
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with at least 50% reduction in Anti-beta2-glycoprotein test Immunoglobulin G (abeta2GPI IgG) levels | At week 48 compared to week 0
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with a negative Lupus Anticoagulant (LA) test | At weeks 4, 9, 12, 18, 24, 36 and 48
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with a negative Lupus Anticoagulant (LA) test | At week 24
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method
Change in Anti-beta2-glycoprotein test Immunoglobulin G (abeta2GPI IgG) levels | From weeks 0 to weeks 4, 9, 12, 18, 24, 36 and 48
  Fold-change from week 0 will be summarized within dosing cohort using descriptive statistics. Additional descriptive statistics may include absolute change and ordinal definitions of antibody levels
Change in Anticardiolipin antibodies Immunoglobulin M (aCL IgM) levels | From week 0 to weeks 4, 9, 12, 18, 24, 36 and 48
  Fold-change from week 0 will be summarized within dosing cohort using descriptive statistics. Additional descriptive statistics may include absolute change and ordinal definitions of antibody levels
The proportion of Grade 2 or higher serious adverse event (SAEs) related to daratumumab | At or before weeks 9, 24, and 48
  The proportion of participants who experience at least one event will be estimated by dosing level with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with at least 50% reduction in Anti-beta2-glycoprotein I antibodies (a-beta2GPI IgG) compared to week 0 | At week 9
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with a negative Lupus Anticoagulant (LA) test | At week 48
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method
The proportion of participants with at least 50% reduction in Anticardiolipin antibodies Immunoglobulin G (aCL IgG) levels | At week 48 compared to week 0
  For dichotomous endpoints, including the composite of (a) Negative LA test, and (b) fold-reduction in both aCL IgG and aß2GPI IgG, and the individual components, proportions will be reported with 90% confidence intervals derived using the Clopper-Pearson exact method

CONTACTS AND LOCATIONS:
Overall Officials: Doruk Erkan, M.D., M.P.H., Study Chair — Hospital for Special Surgery, New York: Division of Rheumatology; Jason Knight, M.D., Ph.D., Study Chair — University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology
Locations (8):
- United States (8):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Northwell Health, Great Neck, New York
  - NYU Langone, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Weill Cornell, New York, New York
  - Duke University, Durham, North Carolina

REFERENCES:
- See also: Immune Tolerance Network — https://www.immunetolerance.org/
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait